CLINICAL TRIAL: NCT00270738
Title: Treatment for Stress Urinary Incontinence-Indirect Training of Pelvic Floor Muscle Via Transversus Abdominis Muscle Contraction
Brief Title: Treatment for Female Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9461700665
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Female Urinary Incontinence
Keywords: urinary incontinence; transversus abdominis; pelvic floor muscles; randomized controlled trial
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): TrA training group
  Interventions: Procedure: Indirect training of the PFMs via transversus abdominis
- 2 (Active Comparator): PFMT group
  Interventions: Procedure: pelvic floor muscle training
- 3 (Active Comparator): control group (PFM exercise at home)
  Interventions: Procedure: home exercise

INTERVENTIONS:
Procedure: Indirect training of the PFMs via transversus abdominis — Individual visit: twice a month for 4 months. Exercise regimen: diaphragmatic breathing, tonic activation, muscle strengthening, functional expiratory patterns, and impact activities.
  Other Names: TrA training
  Arms: 1
Procedure: pelvic floor muscle training — Individual visit: twice a month for 4 months. Exercise: intensive pelvic floor muscle training
  Other Names: PFMT
  Arms: 2
Procedure: home exercise — PFM exercise at home: at least six high-intensity (near-maximum) contractions 3 times per day at home, with an aim at holding each muscle contraction for 10 seconds, with at least a 10-second rest between contractions.
  Arms: 3

SUMMARY:
Urinary incontinence (UI) is the complaint of any involuntary leakage of urine. Stress urinary incontinence (SUI) is the complaint of involuntary leakage on effort or exertion, or on sneezing or coughing. The prevalence of female UI is greater than that of male, and the commonest type is SUI. UI has significant impact on the quality of life including physical, mental and social issues. SUI may also lead to withdraw from regular physical exercise and fitness activities that important in the prevention of osteoporosis, coronary heart disease, and so on. The cause of SUI is related to the impairment of pelvic floor muscles (PFM). So far, the effects of intensive pelvic floor muscle training for female SUI were proved in many randomized controlled trials. However, training of accurate contraction of PFM depends on vaginal palpation. The willingness to seek for medical help may be reduced due to being embarrassed with vaginal palpation. Sapsford proposed a concept to treat SUI via transversus abdominis (TrA) that does not need to palpate the vagina. Maybe the new intervention can promote the willingness to seek medical help. However, to date there is no randomized controlled trial comparing the effect of indirect training of the PFM via TrA with either untreated control or other intervention. Therefore, there are two purposes in this study, to compare the effect of indirect training of PFM via TrA with control group and to compare the effect of indirect training of PFM via TrA with PFMT for female SUI.

DETAILED DESCRIPTION:
In the first period (part I), 100 women with SUI will be recruited in this study and randomized to intervention or control group after stratified by the moving direction of PFM during contraction of TrA. All subjects will be evaluated pre- and post- 4-month intervention. The measurements included basic data and comprehensive urogynaecological history, women's observations, quantification of symptoms, clinician's measures and quality of life.

Women in the control group will receive customary information of PFM exercise and they can decide by themselves to receive an intensive pelvic floor muscle training after control period or not. The intervention group will follow a specially designed exercise course including diaphragmatic breathing, tonic activation, muscle strengthening, functional expiratory patterns and impact activities. They will be individually trained by a physical therapist for 30-60 minutes eight times during intervention period.

In the second period (part II), another 100 women with SUI will be recruited in this study and randomized to intervention or control group. All subjects will be evaluated pre- and post- 4-month intervention. The measurements included basic data and comprehensive urogynaecological history, women's observations, quantification of symptoms, clinician's measures and quality of life.

Women in the control group will receive customary information of PFM exercise and they can decide by themselves to receive intensive pelvic floor muscle training after control period or not. The intervention group will received intensive pelvic floor muscle training. They will be individually trained by a physical therapist for 30-60 minutes eight times during intervention period.

Descriptive and inferential statistics will be completed using SPSS for windows, version 11.0. Descriptive statistics will be computed for subject demographics. Normality will be evaluated by using the Shapiro-Wilk test for all variables. The confounding factors between two groups will be tested by the independent t-test or Chi-square test. A two-way mixed analysis of variance (ANOVA) and Friedman test will be used to assess possible difference between pre- and post- intervention and two groups. The Chi-square will be used to assess the discount dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* female with stress urinary incontinence episodes during last month

Exclusion Criteria:

* Systemic neuromuscular disease
* Previous medication、surgery、PFMT for urinary incontinence
* Previous surgery of bladder or low back
* RAH
* During pregnancy or after childbirth<3 m/o
* Severe prolapse of bladder or uterus

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
women's observations | 4 months

SECONDARY OUTCOMES:
quantification of symptoms | 4 months
clinical measures | 4 months
quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Study Director — Graduate School of Physical Therapy, College of Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hung HC, Chih SY, Lin HH, Tsauo JY. Exercise adherence to pelvic floor muscle strengthening is not a significant predictor of symptom reduction for women with urinary incontinence. Arch Phys Med Rehabil. 2012 Oct;93(10):1795-800. doi: 10.1016/j.apmr.2012.03.010. Epub 2012 Mar 23. PMID 22446154
- [Derived] Hung HC, Hsiao SM, Chih SY, Lin HH, Tsauo JY. Effect of pelvic-floor muscle strengthening on bladder neck mobility: a clinical trial. Phys Ther. 2011 Jul;91(7):1030-8. doi: 10.2522/ptj.20100186. Epub 2011 May 12. PMID 21566065